CLINICAL TRIAL: NCT04091841
Title: The Effect of Protein Supplement on Vertebral Fusion and Enhanced Recovery After Posterior Spine Fusion Surgery
Brief Title: Trial of Protein Supplement on Vertebral Fusion in Posterior Spine Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Principal Investigator, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1398/022
Record Dates: First submitted 2019-08-05; First posted 2019-09-17 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Spine Surgery
Keywords: Protein supplement; Protein diet; Vertebral fusion; Enhanced recovery after surgery; Infection; Wound healing; Pain
MeSH Terms: conditions — Infections; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protein supplement (Experimental): Intervention patients will be received protein diet (1.2 g/kg/day) and protein supplement (36 g/day) for 1 month after surgery.
  Interventions: Drug: protein supplement
- Carbo Mass (Placebo Comparator): Control patients will be received protein diet (1.2 g/kg/day) and Carbo Mass for 1 month after surgery.
  Interventions: Other: Carbo Mass

INTERVENTIONS:
Drug: protein supplement — Three sachet of protein supplement to be mixed in with water used daily.
  Other Names: Pure-protein
  Arms: protein supplement
Other: Carbo Mass — Three sachet of Carbo Mass supplement to be mixed in with water used daily.
  Arms: Carbo Mass

SUMMARY:
Receiving protein can affect the bone formation and maintenance by providing a structural matrix of the bone, optimizing the level of IGF-1, increasing intestinal calcium absorption, transferring phosphorous, and improving muscle strength.Therefore, protein may be effective on vertebral fusion by such mechanisms. In this trial patients undergoing elective posterior spine fusion surgery are divided into two groups of intervention or control.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in patients undergoing elective posterior spine fusion surgery in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. The participants are 80 eligible posterior spine fusion surgery patients, aged ≥ 18 years. Intervention patients will be received 36 grams of protein supplement along with diet containing 1.2 g/kg/day of protein for 30 days after surgery and control patients will be received Carbo Mass along with diet containing 1.2 g/kg/day of protein 30 days after surgery. Patients will be evaluated for occurrence of vertebral fusion and enhanced recovery after 3 months surgery.

ELIGIBILITY:
Inclusion criteria:

* Adult patients 18-65 years
* Body mass index 18.5-30
* Candidate for the elective posterior spine fusion
* Without history of severe liver disorder
* Without history of Kidney disorder
* Without history of diabetes
* Without history of trauma and fracture of the vertebral
* Without history of osteoporosis
* Without history of Gastrointestinal malabsorption
* Without history of Parathyroid gland disorders
* Without taking medications that affect the metabolism of bone, such as calcitonin,
* bisphosphonate, corticosteroid
* No smoking
* serum level of vitamin 25 (OH) D ≤20 ng/l

Exclusion Criteria:

* Allergy or intolerance to protein or maltodextrine supplement
* Unwillingness to continue cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of vertebral fusion in CT scan | 6 months after surgery
  Rate of formation of a solid bony Union in CT scan

SECONDARY OUTCOMES:
Rate of wound healing | Discharge, 15 days and 1 month after surgery
  Rate of wound healing, the sutures of the surgery, inspected by granulation tissue formation.
Rate of of wound infection | 15 days, 1 and 3 month after surgery
  Rate of of wound infection, revealed by physical examination
score of pre and postoperative pain | baseline, discharge, 15 days 1 and 3 month after surgery
  pain measured by the visual analogue scale or visual analog scale (VAS) questionnaire
Concentration of serum IGF-1 | baseline, 1 month after surgery
  Concentration of Insulin-like growth factor-1
Concentration of serum albumin | baseline, 1 month after surgery
  Concentration of serum albumin
Concentration of serum total protein | baseline, 1 month after surgery
  Concentration of serum total protein
Concentration of serum hsCRP | baseline, 48 hour,15 days and 1 month after the surgery
  Concentration of serum high-sensitivity C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: zahra vahdat shariatpanahi, MD,PhD, Study Chair — Faculty of Nutrition and Food Technology, SBMU
Locations (1):
- Zahra vahdat shariatpanahi, Tehran, Iran